CLINICAL TRIAL: NCT02101359
Title: Efficacy and Safety Assessment of Intracameral Injection of T2380 in Cataract Surgery Versus Reference Group (Topical Mydriatics and Anaesthetic)
Brief Title: Efficacy and Safety Assessment of Intracameral Injection of T2380 in Cataract Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratoires Thea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LT2380-PIII-05/10
Record Dates: First submitted 2013-09-04; First posted 2014-04-02 (Estimated); Results first posted 2014-09-25 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Mydriatics; Tropicamide; Tetracaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- T2380 (Experimental): Topical anaesthetic: Tetracaine was instilled in the eye to be operated before surgery.
  At the beginning of surgery, 200 μL of T2380 were administrated intracamerally.
  Interventions: Drug: T2380; Drug: Tetracaine
- Mydriatics and anesthetic (Active Comparator): Topical anaesthetic: Tetracaine was instilled in the eye to be operated before surgery.
  Topical Mydriatic treatments were instilled three times before surgery.
  Interventions: Drug: Mydriatics; Drug: Tetracaine

INTERVENTIONS:
Drug: T2380 — 200 microlitres of T2380 will be administrated intracamerally
  Arms: T2380
Drug: Mydriatics — 3 drops of tropicamide and phenylephrine were instilled 30 minutes before surgery. The second and the third instillation of both phenylephrine and tropicamide will be realised respectively within 20 and 10 minutes before surgery.
  Other Names: Tropicamide, Phenylpehrine
  Arms: Mydriatics and anesthetic
Drug: Tetracaine — Two drops of tetracaine were instilled in the eye to be operated 5 minutes and 1 minute before surgery
  Other Names: Tetracaine 1%

SUMMARY:
The purpose of this study is to determine the efficacy and safety assessment of T2380 for mydriasis and anaesthesia in phacoemulsification cataract surgery versus reference group (topical mydriatics and anaesthetic) 2X246 patients.

DETAILED DESCRIPTION:
In order to perform pupil size measurements and ocular discomfort assessments at specific times, the surgical procedure was divided into 5 time periods according to the following time points: T1 (just before first incision), T2 (just before viscoelastic injection), T3 (just before capsulorhexis), T4 (just before intraocular lens injection), and T5 (just before cefuroxime injection).

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent
* Male or female aged from 40 to 88 years old
* Scheduled to undergo unilateral cataract surgery

Exclusion criteria:

* Combined surgery
* Previous intraocular surgery

Ages: 40 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 609 (Actual)
Dates: Start 2011-06; Primary Completion 2013-01 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph COLIN, Principal Investigator; Marc LABETOULLE, Principal Investigator
Locations (1):
- Laboratoires Thea, Clermont-Ferrand, France

REFERENCES:
- [Derived] Labetoulle M, Behndig A, Tassignon MJ, Nuijts R, Mencucci R, Guell JL, Pleyer U, Szaflik J, Rosen P, Berard A, Chiambaretta F, Cochener-Lamard B; Intracameral Mydrane (ICMA), Ethics Group. Safety and efficacy of a standardized intracameral combination of mydriatics and anesthetic for cataract surgery in type-2 diabetic patients. BMC Ophthalmol. 2020 Mar 3;20(1):81. doi: 10.1186/s12886-020-01343-x. PMID 32126990
- [Derived] Labetoulle M, Findl O, Malecaze F, Alio J, Cochener B, Lobo C, Lazreg S, Hartani D, Colin J, Tassignon MJ, Behndig A; Intracameral Mydrane Study 2 Group. Evaluation of the efficacy and safety of a standardised intracameral combination of mydriatics and anaesthetics for cataract surgery. Br J Ophthalmol. 2016 Jul;100(7):976-985. doi: 10.1136/bjophthalmol-2015-307587. Epub 2015 Nov 3. PMID 26531052

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The patients, fulfilling the criteria for inclusion were invited to participate in the study.
Groups:
- T2380: T2380: Intracameral administration during surgery
- Reference Group: Mydriatics and anesthetics: Topical treatments used the day of surgery
Period: Overall Study
Arm/Group | T2380 | Reference Group
Started | 295 | 296
Completed | 266 | 277
Not Completed | 29 | 19
Not completed — Not included | 23 | 13
Not completed — Withdrawal by Subject | 5 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 0 | 2

BASELINE CHARACTERISTICS:
Population: 609 patients have signed the informed consent, but 18 patients were not selected and /or not randomised.
  591 patients were randomised (at selection visit).
Groups:
- Reference Group: Mydriatics and anesthetic: Topical treatments used the day of surgery
- Total: Total of all reporting groups
Arm/Group | T2380 | Reference Group | Total
Number analyzed (Participants) | 295 | 296 | 591
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.2 (9.4) | 70.6 (9.2) | 69.9 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120 | 134 | 254
  Male | 175 | 162 | 337
Region of Enrollment [Number; unit: participants]
  Algeria | 32 | 31 | 63
  Austria | 11 | 10 | 21
  Belgium | 17 | 16 | 33
  France | 192 | 188 | 380
  Germany | 9 | 8 | 17
  Italy | 11 | 11 | 22
  Spain | 6 | 11 | 17
  Sweden | 9 | 9 | 18
  Portugal | 8 | 12 | 20

OUTCOME MEASURES:

1. Primary Outcome: The Primary Efficacy Variable is Response Based on the Realisation of the Capsulorhexis Without Use of Any Additive Mydriatic Treatment.
Time Frame: Day 0
Population: Modified ITT (mITT) Set: All randomised patients for whom there was evidence they used the study medication, and who satisfied the non-inclusion criterion concerning unauthorized previous and concomitant medications. Patients were assigned to the treatment group as treated.
Measure: Number; unit: percentage of responders
Arm/Group | T2380 | Reference Group
Number analyzed (Participants) | 268 | 281
percentage of responders | 98.9 | 94.7

ADVERSE EVENTS:
Arm/Group | T2380 | Reference Group
Serious Adverse Events (participants affected / at risk) | 4/295 | 6/296
Other Adverse Events (participants affected / at risk) | 0/295 | 0/296
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | T2380 (N=295) | Reference Group (N=296)
Macular oedema (Eye disorders) | 1 | 0
Keratitis (Eye disorders) | 1 | 0
Cataract operation complication (Injury, poisoning and procedural complications) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Eye haemorrhage (Eye disorders) | 0 | 1
Retinal detachment (Eye disorders) | 0 | 1
Posterior capsule rupture (Eye disorders) | 0 | 1
Vascular bypass dysfunction (Injury, poisoning and procedural complications) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All the results of the Trial are the sole and exclusive property of THEA, and cannot be used in whatever form without prior written agreement of THEA.